CLINICAL TRIAL: NCT00006202
Title: Dose Ranging Study of Lutein Supplementation in Persons Over Age 60
Brief Title: Lutein for Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000208; 00-EI-0208
Record Dates: First submitted 2000-09-09; First posted 2000-09-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: Macular Degeneration
Keywords: Serum levels of Lutein; Age-Related Macular Degeneration; Safety; Toxicity
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein

INTERVENTIONS:
Drug: Lutein

SUMMARY:
This study will examine whether taking the vitamin lutein changes lutein blood levels. Lutein, vitamin C, vitamin E and beta-carotene may be useful in treating the eye disease age-related macular degeneration, but more information is needed to support this. Age-related macular degeneration can significantly impair the ability to read, drive, and carry out daily activities. It is the most common cause of vision loss in people over age 60. Lutein a carotenoid that occurs naturally in the retina (the back part of the eye), especially the macula-the part of the retina that is important for fine, detailed vision.

Men and women 60 years of age and older, with or without age-related macular degeneration, may be eligible for this study. Candidates will undergo the following tests:

1. Medical history and physical examination.
2. Eye examination-Includes evaluation of visual acuity, measurement of eye pressure, examination of the lens, retina, pupils and eye movements, and photographs of the eye.
3. Visual field study-Examines the ability to see objects in the periphery. The subject looks at a target on a screen and indicates when lights that appear in other places on the screen are visible.
4. Flicker photometry-The subject looks at a flashing light and turns a knob until the light stops flashing.
5. Blood tests-To measure blood levels of lutein and other carotenoids, liver function, cholesterol and triglycerides.

Participants will be randomly assigned to take one of three dosages of lutein (2.5 milligrams, 5 milligrams or 10 milligrams) for 6 months and will be examined at follow-up visits scheduled 1, 3, 6, 9 and 12 months after starting lutein. During these visits, many of the exams described above will be repeated to evaluate the effects of lutein treatment on the eye.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the association of varying doses of oral supplementation of lutein with the resulting serum levels of lutein in people over age 60 who may or may not have AMD. Secondary objectives are to investigate the relationship between level of disease and lutein absorption and to assess change in macular pigment. Assessment of macular pigment is not routinely performed in this patient population. Including this assessment in the current study will further attempts to standardize its implementation. If results appear to warrant further study, a placebo-controlled study may be appropriate. Patients will range from those with no AMD and little or no drusen in either eye through end stage AMD (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in the eye with worst disease. AMD severity will be classified using Age-Related Eye Disease Study criteria for the definition of advanced AMD (Appendix 2). Development of a safety profile is not a specific objective of this study. To this point in time, the available published data have not indicated any safety concerns. However, due to the lack of complete knowledge of potential toxicities, safety assessments will be performed at all scheduled study visits. These safety assessments include: visual acuity, complete ophthalmic examination, fundus photos, liver function tests, visual field tests, and a side-effect questionnaire from the AREDS. Should safety concerns arise, adverse event rates can be compared to the AREDS, which is based on the same study population.

ELIGIBILITY:
INCLUSION CRITERIA:

Men and women aged 60 years or older.

Patients ranging from no AMD with little or no drusen in either eye through end stage AMD (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in their eye with worst disease will be eligible.

The ability to understand and sign an informed consent form prior to enrollment.

EXCLUSION CRITERIA:

Ocular disease which confounds assessment of the retina other than age-related macular degeneration including diabetic retinopathy, central serous choroidopathy, optic atrophy, retinal vein occlusion, active uveitis, significant explained or unexplained visual field loss, or any other type of retinopathy or retinal degeneration.

Chronic requirement for any systemic or ocular medication for other diseases such as glaucoma.

Patients has regularly been taking lutein supplements during the last 3 months or is currently taking lutein supplements. The daily use of the new Centrum or Centrum Silver or other similar multivitamins will be allowed but should be limited to a maximum of twice a day.

Abnormal liver function tests.

Inability to be followed for a period of 1 year.

Acute potentially life-threatening illness such as heart attack in the last year, malignant cancer or blood disease not in remission.

History of lung cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2000-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Machemer R, Steinhorst UH. Retinal separation, retinotomy, and macular relocation: II. A surgical approach for age-related macular degeneration? Graefes Arch Clin Exp Ophthalmol. 1993 Nov;231(11):635-41. doi: 10.1007/BF00921957. PMID 8258397
- [Background] de Juan E Jr, Loewenstein A, Bressler NM, Alexander J. Translocation of the retina for management of subfoveal choroidal neovascularization II: a preliminary report in humans. Am J Ophthalmol. 1998 May;125(5):635-46. doi: 10.1016/s0002-9394(98)00018-x. PMID 9625547
- [Background] Seddon JM, Ajani UA, Sperduto RD, Hiller R, Blair N, Burton TC, Farber MD, Gragoudas ES, Haller J, Miller DT, et al. Dietary carotenoids, vitamins A, C, and E, and advanced age-related macular degeneration. Eye Disease Case-Control Study Group. JAMA. 1994 Nov 9;272(18):1413-20. PMID 7933422
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300